CLINICAL TRIAL: NCT02303639
Title: Medical ANtiarrhythmic Treatment or Radiofrequency Ablation in Ischemic Ventricular Tachyarrhythmias. A Prospective, Randomized Multicentre Study.
Brief Title: Medical ANtiarrhythmic Treatment or Radiofrequency Ablation in Ischemic Ventricular Tachyarrhythmias
Acronym: MANTRA-VT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Finland Hospital District (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7U/2014
Record Dates: First submitted 2014-11-21; First posted 2014-12-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Myocardial Infarction; Ventricular Tachyarrhythmia
Keywords: implantable cardioverter defibrillator; antiarrhythmic medication; catheter ablation
MeSH Terms: conditions — Myocardial Infarction; Tachycardia, Ventricular | interventions — Catheter Ablation; Amiodarone; Sotalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiofrequency catheter ablation (Experimental): Radiofrequency catheter ablation using open-irrigated ablation catheter and 3D electroanatomical mapping
  Interventions: Procedure: Radiofrequency catheter ablation
- Antiarrhythmic drug therapy (Active Comparator): Amiodarone (or sotalol) tablet by mouth for the duration of the study
  Interventions: Drug: Antiarrhythmic drug therapy

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation — Catheter ablation with an open-irrigated tip ablation catheter and 3D electroanatomical mapping
  Arms: Radiofrequency catheter ablation
Drug: Antiarrhythmic drug therapy — Amiodarone (or sotalol) for prevention of VT/VF relapses
  Other Names: amiodarone; sotalol; class III antiarrhyhtmic agents
  Arms: Antiarrhythmic drug therapy

SUMMARY:
The study evaluates whether catheter based radiofrequency ablation is superior to optimized antiarrhythmic medical therapy in preventing ventricular tachyarrhythmia relapses in patients with ischemic heart disease and implantable cardioverter defibrillator.

DETAILED DESCRIPTION:
The study is designed to evaluate whether catheter based radiofrequency ablation is superior to optimized antiarrhythmic medical therapy in preventing ventricular tachyarrhythmia relapses among patients with prior myocardial infarction and implantable cardioverter defibrillator (ICD). The patients have not been using using chronic antiarrhythmic medication. Primary end point is number of ICD therapies (defibrillations, cardioversions and antitachycardia pacing) and otherwise documented sustained ventricular tachycardia (duration more than 30 s or hemodynamically unstable ) or ventricular fibrillation episodes during 12 months follow-up period. Secondary end points include mortality, hospitalization for cardiac reason, health economics, quality of life and several ICD and arrhythmia related issues. Total length of the follow-up is at least two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years of age with prior myocardial infarction and ICD (single chamber, dual chamber ICD or ICD with biventricular pacing capability (CRT-D)) for primary or secondary prevention of sudden cardiac death (SCD), who have had at least two documented episodes of sustained VT or VF and no chronic amiodarone treatment for ventricular tachyarrhythmias

Exclusion Criteria:

* Age less than 18 years or more than 80 years
* Non-ischemic cardiomyopathy
* Ongoing chronic treatment of ventricular tachyarrhythmias with amiodarone, intolerance/contraindication to all class III antiarrhythmic drugs (i.e., intolerance/contraindication to one class III agents is not excluding the patient if another one can be used)
* Contraindication to endocardial catheter ablation (e.g., intracavitary thrombi, contraindication to perioperative anticoagulation)
* Previous VT/VF ablation
* Open heart surgery within 3 months
* Prosthetic heart valve
* Planned revascularization (PCI or CABG)
* Surgery for structural heart disease or heart transplantation
* Pregnancy or planned pregnancy within the follow-up period
* Secondary cause for VT/VF (e.g., acute myocardial infarction)
* Patient does not want to participate
* Life expectancy less than 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of ventricular tachycardia (VT) or ventricular fibrillation (VF) episodes | 12 months
  • Number of appropriate ICD therapies (defibrillation, cardioversion, antitachycardia pacing) for VT/VF and otherwise documented sustained VT or VF episodes at 12 months

SECONDARY OUTCOMES:
All cause mortality | 12 and 24 months
Cardiovascular mortality | 12 and 24 months
Time to first hospitalization and number of hospital days | 12 and 24 months
Comparative cost-effectiveness of the therapies | 12 and 24 months
Quality of life measured By SF-36 and EQ5D questionnaires | 12 and 24 months
Patient related outcome measured by the PHQ-9, GAD-7, ICDC-8 and EXPECT-ICD questionnaires | 12 and 24 months
Number of appropriate ICD therapies and sustained VT/VF episodes | 24 months
Number of non-sustained VT episodes | 12 and 24 months
Number of electrical storm episodes | 12 and 24 months
Time to first VT/VF | up to 24 months
Time to reablation | up to 24 months
Number of inappropriate ICD therapies | up to 24 months
Number of atrial fibrillation and other supraventricular arrhythmia episodes | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Raatikainen, MD PhD, Principal Investigator — Keski-Suomen sairaanhoitopiiri
Locations (2):
- Finland (2):
  - Central Finland Central Hospital, Jyväskylä
  - Heart Center Tampere University Hospital, Tampere